CLINICAL TRIAL: NCT04236297
Title: Evaluation of Modified Bite-Block vs Standard Bite Block for Invasive Imaging Procedures
Brief Title: Evaluation of Modified Bite-Block for Invasive Imaging Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Srdjan Jelacic, Assistant Professor, School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004883
Record Dates: First submitted 2020-01-10; First posted 2020-01-22 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Bite Block
Keywords: bite block, transesophageal echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Bite Block (Other): Patients undergoing transesophageal echocardiogram under sedation or general anesthesia during which a modified bite block is used
  Interventions: Device: bite block

INTERVENTIONS:
Device: bite block — Physicians performing transesophageal echocardiogram in patients under sedation or general anesthesia will use either standard or modified bite block.

SUMMARY:
The purpose of this study is to compare a modified bite block with standard bite block during transesophageal echocardiography procedures in patients who are either sedated or under general anesthesia.

These dental protector devices are class I devices which are exempt from the FDA 510(k) premarket notification requirements.

DETAILED DESCRIPTION:
Bite block is a single-use medical device used to keep the mouth open during invasive imaging procedures and prevent the patient from biting the imaging probe.

The purpose of this study is to compare a modified bite block with standard bite block during transesophageal echocardiography exam procedures in patients who are either sedated or under general anesthesia.

The commercially available bite blocks are almost exclusively made of hard plastic that does not conform well to the patient's mouth with additional protrusions used to secure the bite block in place that have the potential to cause patient injury. Hard plastic is used to prevent patient from biting down on the imaging probe while side protrusions are used to strap the bite block down to prevent dislodgment.

Modified bite block is made of softer material with improved mouth fit and no need for strapping the bite block to keep it in place. Softer material is more comfortable while the designs mimics mouth guard used in dentistry to protect patient's teeth and keep the bite block in place while sleeping.

The specific aims of this project include:

* assessment of patient comfort during invasive imaging procedure
* assessment of provider satisfaction with the bite block
* assessment of patient lip/gum/teeth injury after bite block use
* assessment of imaging probe damage after procedure
* assessment of bite block's ability to stay in place during procedure

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing stand-alone transesophageal echocardiography exam under sedation or general anesthesia
* Undergoing procedure that requires transesophageal echocardiography exam during the procedure under general anesthesia
* Cardiology and cardiac anesthesiology echocardiographers performing transesophageal echocardiography exam who wish to participate

Exclusion Criteria:

* Less than 18 years of age
* Any procedure that does not require transesophageal echocardiography exam during the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Oral injury | Within 24 hours
  Number of participants with oral injury (dental injury, lacerations/bruises on gums and lips) which will be determined by examination

SECONDARY OUTCOMES:
Dislodgment | Within 24 hours
  Number of participants with bite block dislodgment which will be determined by provider questionnaire
Provider satisfaction | Within 24 hours
  Number of providers that would use standard or redesigned bite block again

CONTACTS AND LOCATIONS:
Overall Officials: Srdjan Jelacic, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No